CLINICAL TRIAL: NCT03939806
Title: Renal Effects of Carbetocin and Oxytocin in Cesarean Section for Preventing Post-partum Haemorrhage: a Prospective Randomized Study
Brief Title: Effects of Oxytocin and Carbetocin on Renal System in Cesarean Sections
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Gamze Sinem Caglar, Clinical Professor, Ufuk University
Other Study IDs: CO2019
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; carbetocin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Oxytocin: This group will be given 3 IU / 3 ml oxytocin (intravenously) after the clamping of the umbilical cord. Uterine tonus will be assessed after 60 seconds and if it is lower than 7, oxytocin 3 IU / 3 ml will be repeated, up to a maximum of three times. If uterine tonus is still lower than 7, rescue uterotonics such as intramuscular methylergonovine or intravenous misoprostol will be administered.
  Interventions: Drug: Oxytocin
- Carbetocin: This group will be given 100 mcg / 3 ml carbetocin (intravenously) after the clamping of the umbilical cord. If uterine tonus is lower than 7, rescue uterotonics such as intramuscular methylergonovine or intravenous misoprostol will be administered.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Oxytocin — To be given to Oxytocin group following the clamping of the umbilical cord
  Groups: Oxytocin
Drug: Carbetocin — To be given to Carbetocin group following the clamping of the umbilical cord
  Groups: Carbetocin

SUMMARY:
The aim of this study is to evaluate the renal outcome of patients undergoing elective C/S where oxytocin or carbetocin is used for postpartum hemorrhage prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Term (>37 weeks of gestation) uncomplicated pregnant women undergoing elective cesarean section

Exclusion Criteria:

* Patients refusing to participate in the study
* Complicated pregnancies
* Patients with risk factors for postpartum hemorrhage
* Contraindications for oxytocin or carbetocin usage
* Patients with known renal diseases
* Preterm births (<37 weeks of gestation)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population consists of term (gestational age greater than 37 weeks) pregnant women scheduled to undergo elective cesarean section.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Urine volume | Intraoperative period
  Total amount of intraoperative urine output in milliliters
Urinary sodium | Preoperative, Postoperative 2nd, 4th, 24th hours
  The change in urinary sodium content (milligrams) compared to the preoperative period
Blood sodium | Preoperative, Postoperative 2nd, 4th, 24th hours
  The change in blood sodium content (milligrams) compared to the preoperative period

SECONDARY OUTCOMES:
Blood osmolality | Preoperative, Postoperative 2nd, 4th, 24th hours
  The change in blood osmolality compared to the preoperative period
Blood loss | Intraoperative period
  The total volume of intraoperative blood loss
Need for additional uterotonics | Starting from the preoperative period, ending at the 24th postoperative hour
  Total dose (milligrams) of additional uterotonics administered
Blood transfusion | Starting from the clamping of the umbilical cord, ending at the 24th postoperative hour
  Total volume (milliliters) of blood transfused

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University Faculty of Medicine Hospital, Ankara, Balgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larciprete G, Montagnoli C, Frigo M, Panetta V, Todde C, Zuppani B, Centonze C, Bompiani A, Malandrenis I, Cirese A, Valensise H. Carbetocin versus oxytocin in caesarean section with high risk of post-partum haemorrhage. J Prenat Med. 2013 Jan;7(1):12-8. PMID 23741542
- [Background] Engstrom T, Barth T, Melin P, Vilhardt H. Oxytocin receptor binding and uterotonic activity of carbetocin and its metabolites following enzymatic degradation. Eur J Pharmacol. 1998 Aug 21;355(2-3):203-10. doi: 10.1016/s0014-2999(98)00513-5. PMID 9760035